CLINICAL TRIAL: NCT07395505
Title: From Cure to Quality: Advancing Surgical and Postoperative Outcomes in Pelvic Exenteration
Brief Title: Postoperative Results and Outcomes in Surgical Pelvic Exenteration
Acronym: PROS-PE
Status: Enrolling by invitation | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202501190A3C5001
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer Recurrent; Pelvic Exenteration; Advanced Rectal Cancer
Keywords: Advanced rectal cancer; Recurrent rectal cancer; Pelvic exenteration; Sacrectomy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic Exenteration Group: Adult patients with locally advanced or recurrent rectal adenocarcinoma invading adjacent organs undergo pelvic exenteration under a standardized multidisciplinary surgical protocol.

SUMMARY:
The purpose of this study is to evaluate the feasibility of a standardized surgical and care process for patients with locally advanced or recurrent rectal cancer that has spread to nearby pelvic organs. When cancer invades adjacent structures (such as the sacrum, bladder, or prostate), a complex procedure called pelvic exenteration (PE) is often required to remove the tumor entirely.

This research does not involve testing new or experimental surgical techniques. All procedures performed in this study are part of standard clinical practice. Instead, the focus of this project is to:

Standardize Procedures: Create consistent, high-quality steps for the surgical team to follow.

Improve Teamwork: Enhance coordination between different medical specialists (such as colorectal surgeons, urologists, and oncologists) to provide better care.

Track Outcomes: Use a patient registry to monitor clinical data and quality of life after surgery through patient-reported surveys.

A total of 24 adult patients will be enrolled over a three-year period. By refining these workflows and monitoring patient recovery, the study aims to ensure that these complex surgeries are performed as safely and effectively as possible.

DETAILED DESCRIPTION:
This prospective, single-center surgical feasibility study is designed to establish and validate standardized protocols for patients undergoing pelvic exenteration (PE), with or without sacrectomy, for locally advanced or recurrent rectal cancer invading adjacent pelvic structures.

The study focuses on three primary operational pillars:

1. Standardization of Surgical Techniques and SOPs The project aims to refine and standardize complex surgical maneuvers to ensure technical consistency across cases. This includes:

   Precise identification and preservation of pelvic nerves.

   Intraoperative assessment of sacrectomy levels (specifically targeting S2-S4).

   Standardization of urological procedures and advanced reconstructive approaches for the pelvic floor.

   Implementation and practical validation of Standard Operating Procedures (SOPs) to achieve consistent R0 resection margins.
2. Prospective Data Integration and Quality of Life Monitoring A systematic case registry will be established to capture comprehensive perioperative clinical data. Beyond clinical metrics, the study integrates Patient-Reported Outcome Measures (PROMs) to evaluate the impact of PE on long-term postoperative function and quality of life. This data will be used to optimize clinical workflows and improve patient counseling regarding functional recovery.
3. Multidisciplinary Team (MDT) Synergy The study reinforces a collaborative care model involving colorectal surgery, urology, orthopedics, oncology, radiology, and pathology. By strengthening MDT collaboration, the project aims to enhance perioperative care quality, from preoperative surgical candidacy review to postoperative management.

As a feasibility study, the enrollment of 24 patients over three years will serve as a pilot to confirm the practicality of these SOPs and the efficiency of the MDT workflow in a high-complexity surgical setting. All procedures fall within the scope of standard clinical practice; the research focus remains on the optimization of care delivery and process standardization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥20 years.
* Histologically confirmed rectal adenocarcinoma or anal adenocarcinoma.
* Tumor invasion of sacrum (requiring sacrectomy, S2-S4) or anterior structures (e.g., prostate), or lateral structures(SLAM, vessels, nerve) where resection of the invaded organ is necessary to achieve R0 resection, as determined by MDT.
* Surgical candidacy confirmed by multidisciplinary review (colorectal surgery, urology, orthopedics, oncology, radiology, pathology).
* Preoperative imaging (MRI, PET/CT) confirming resectable disease without distant metastasis.
* Signed informed consent obtained.

Exclusion Criteria:

* Unresectable disease or widespread distant metastasis.
* Severe comorbidities rendering major surgery or anesthesia unsafe.
* Patients unable to complete postoperative follow-up or unwilling to participate in PROMs assessment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age ≥ 20 years) with histologically confirmed locally advanced or recurrent rectal or anal adenocarcinoma invading adjacent pelvic structures (such as the sacrum, prostate, or bladder) who undergo pelvic exenteration (PE) with or without sacrectomy at Chang Gung Memorial Hospital during the three-year study period.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Short-term outcome | 2026 to 2031
  R0 resection rate
Short-term outcome | 2026 to 2031
  Major complication rate (Clavien-Dindo ≥ III)

SECONDARY OUTCOMES:
Short-term outcome | 2026 to 2031
  Length of stay
Short-term outcome | 2026 to 2031
  readmission rate
Short-term outcome | 2026 to 2031
  90-day mortality

OTHER OUTCOMES:
PROMs：Quality of Life Measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | From recruitment to study completion (approximately 5 years, 2026-2031)
  The EORTC QLQ-C30 is a 30-item questionnaire used to assess the quality of life of cancer patients. Scores are transformed to a scale from 0 to 100. For the functional scales and global health status, higher scores represent a higher (better) level of functioning or quality of life. For the symptom scales, higher scores represent a higher (worse) level of symptoms.
PROMs：Quality of Life Measured by EORTC Quality of Life Questionnaire Colorectal Cancer Module (QLQ-CR29) | From recruitment to study completion (approximately 5 years, 2026-2031)
  This is a 29-item supplemental module specific to colorectal cancer. Scores range from 0 to 100. For functional scales, higher scores indicate better functioning. For symptom scales, higher scores indicate more severe symptoms.
PROMs：Urinary Function Measured by International Prostate Symptom Score (IPSS) | From recruitment to study completion (approximately 5 years, 2026-2031).
  The IPSS consists of 7 questions regarding urinary symptoms and one quality of life question. The total symptom score ranges from 0 to 35. A higher total score indicates a worse outcome (more severe urinary symptoms).
PROMs：Urinary Incontinence Measured by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | From recruitment to study completion (approximately 5 years, 2026-2031).
  The ICIQ-UI SF is a 4-item questionnaire used to evaluate the frequency, severity, and impact of urinary incontinence. The total score ranges from 0 to 21. A higher score indicates a worse outcome (greater severity of urinary incontinence).
PROMs：Male Sexual Function Measured by International Index of Erectile Function (IIEF-5) | From recruitment to study completion (approximately 5 years, 2026-2031).
  The IIEF-5 is a 5-item questionnaire used to evaluate erectile function in male participants. The score ranges from 5 to 25. A higher score represents a better outcome (better erectile function).
PROMs：Female Sexual Function Measured by Female Sexual Function Index (FSFI) | From recruitment to study completion (approximately 5 years, 2026-2031).
  The FSFI is a 19-item questionnaire used to assess sexual function in female participants. The total score ranges from 2 to 36. A higher score represents a better outcome (better sexual function).
PROMs：Bowel Function Measured by Low Anterior Resection Syndrome (LARS) Score | From recruitment to study completion (approximately 5 years, 2026-2031).
  The LARS score is used to assess bowel dysfunction after rectal surgery. The score ranges from 0 to 42. A higher score indicates a worse outcome (more severe bowel dysfunction).
PROMs：Stoma-Related Quality of Life Measured by Stoma Quality of Life (Stoma-QoL) Questionnaire | From recruitment to study completion (approximately 5 years, 2026-2031).
  The Stoma-QoL is a 20-item questionnaire designed to measure quality of life in patients with a stoma. The total score is standardized to range from 0 to 100. A higher score represents a better outcome (better quality of life related to the stoma).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author upon reasonable request

REFERENCES:
- [Result] Hsu YJ, Yu ZH, Jong BK, You JF, Yu YL, Liao CK, Lai CC, Chern YJ. Short- and long-term outcomes of minimally invasive vs. open pelvic exenteration in rectal tumours: a focused meta-analysis. Int J Colorectal Dis. 2025 Apr 3;40(1):86. doi: 10.1007/s00384-025-04876-z. PMID 40180681